CLINICAL TRIAL: NCT05911087
Title: A Phase 2/3, Randomized, Double-blinded , Parallel Controlled Trial to Evaluate the Immunogenicity, Safety and Efficacy of A Heterologous Booster Dose With COVID-19 mRNA Vaccines (Bivalent) , in Previously Vaccinated Subjects Against COVID-19 With 2/3 Doses COVID-19 Vaccine Compared to a Booster Dose With mRNA COVID-19 Vaccine（Pfizer Bivalent Vaccine）in Adults.
Brief Title: A Phase II/III Study to Evaluate the Immunogenicity and Safety and Efficacy of SWIM816 Vaccines for SARS-CoV-2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stemirna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SWP2023-1
Record Dates: First submitted 2023-06-18; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Immunogenicity; Safety

STUDY DESIGN:
Intervention Model Description: randomized#double-blinded # parallel controlled trial#mRNA vaccine# and positive control group#
Who Masked: Participant, Investigator
Masking Description: This study uses an observer-blinded design, and the investigators and participants will all remain blinded before unblinding and do not know which group the participant belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase II group 1 :A single 25 μg dose mRNA vaccine SWIM816 (Experimental): Intervention Name :COVID-19 mRNA vaccine Type :Investigational Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.5ml; Dosage Level(s) :0.25ml; Route of Administration: injection Intramuscular
  Interventions: Biological: Phase II:SWIM816;SARS-Cov-2;
- PhaseII group 2:A single 25 μg dose mRNA vaccine SW-BIC-213 (Active Comparator): Intervention Name :COVID-19 mRNA vaccine Type :Control Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.5ml; Dosage Level(s) :0.25ml; Route of Administration: injection Intramuscular
  Interventions: Biological: Phase II:SW-BIC-213;SARS-Cov-2;
- Phase III group 1:A single 25 μg dose mRNA vaccine SWIM816 (Experimental): Intervention Name :COVID-19 mRNA vaccine Type :Investigational Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.5ml; Dosage Level(s) :0.25ml; Route of Administration: injection Intramuscular
  Interventions: Biological: PhaseIII:SWIM816;SARS-Cov-2;
- Phase III group 2:A single 30 μg dose mRNA Pfizer Bivalent vaccine (Active Comparator): Intervention Name :Pfizer Bivalent Vaccine Type :Control Vaccine Dose :Formulation mRNA Unit Dose Strength(s) :0.3μg; Dosage Level(s) :0.3ml;
  Interventions: Biological: PhaseIII:Pfizer(Pfizer Bivalent vaccine);SARS-Cov-2；

INTERVENTIONS:
Biological: Phase II:SWIM816;SARS-Cov-2; — The study will be performed in people who were previously vaccinated with 2/3 doses of COVID-19 vaccine, with or without previously diagnosed with COVID-19. The interval between the date of last dose and the date of this study vaccination should be 6 to 24 months.
  There are 2 groups in phase 2 stage, total number 200 subjects who are ≥18 years old. Details as below:
  Group 1: (N=100) - SWIM816 25 μg; Group 2: (N=100) - SW-BIC-213 25 μg;
  Arms: Phase II group 1 :A single 25 μg dose mRNA vaccine SWIM816
Biological: Phase II:SW-BIC-213;SARS-Cov-2; — The study will be performed in people who were previously vaccinated with 2/3 doses of COVID-19 vaccine, with or without previously diagnosed with COVID-19. The interval between the date of last dose and the date of this study vaccination should be 6 to 24 months.
  There are 2 groups in phase 2 stage, total number 200 subjects who are ≥18 years old. Details as below:
  Group 1: (N=100) - SWIM816 25 μg; Group 2: (N=100) - SW-BIC-213 25 μg;
  Arms: PhaseII group 2:A single 25 μg dose mRNA vaccine SW-BIC-213
Biological: PhaseIII:SWIM816;SARS-Cov-2; — The study will be performed in people who were previously vaccinated with 2/3 doses of COVID-19 vaccine, with or without previously diagnosed with COVID-19. The interval between the date of last dose and the date of this study vaccination should be 6 to 24 months.
  There are two groups in phase 3 stage., total number 600 subjects who are ≥18 years old. Details as below:
  Group 1: (N=300) - SWIM816 (≥18 years old ) Group 2: (N=300) -Pfizer Bivalent vaccine (≥18 years old)
  Arms: Phase III group 1:A single 25 μg dose mRNA vaccine SWIM816
Biological: PhaseIII:Pfizer(Pfizer Bivalent vaccine);SARS-Cov-2； — The study will be performed in people who were previously vaccinated with 2/3 doses of COVID-19 vaccine, with or without previously diagnosed with COVID-19. The interval between the date of last dose and the date of this study vaccination should be 6 to 24 months.
  There are two groups in phase 3 stage., total number 600 subjects who are ≥18 years old. Details as below:
  Group 1: (N=300) - SWIM816 (≥18 years old ) Group 2: (N=300) -Pfizer Bivalent vaccine (≥18 years old)
  Arms: Phase III group 2:A single 30 μg dose mRNA Pfizer Bivalent vaccine

SUMMARY:
Primary Immunogenicity Objective：Cohort 1: GMTs of SARS-CoV-2 Omicron and related strain neutralizing antibody levels for SWIM816.Cohort 2: To demonstrate the non- inferiority of neutralizing antibody response in terms of geometric mean titers (GMT) of COVID-19 mRNA vaccine(SWIM816) compare with mRNA COVID-19 vaccine(Pfizer Bivalent vaccine) 14 days post dose.

Primary Safety Objective：To assess the reactogenicity and safety of a booster dose in a heterologous vaccination regimen in subjects previously immunized with 2/3 doses of COVID-19 vaccine with or without previously diagnosed with COVID-19.

Secondary Immunogenicity Objectives：To describe the neutralizing antibody response at D29, D91 and D181.To describe binding antibody profile at D01, D15, D29, D91 and D181 of each study group.

Secondary Safety Objective：To assess the reactogenicity and safety of third or fourth booster dose in a heterologous vaccination regimen in subjects previously immunized with 2/3 COVID-19 vaccine doses.

Exploratory Objective：1.Documented confirmed SARS-CoV-2 symptomatic infection；2.Todemonstrate the cellular immune response profile at study group (30 subjects per each group for cellular immune testing).

DETAILED DESCRIPTION:
Endpoints:

Cohorts 1: GMT of SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB) and reference strain neutralizing antibody(Delta and other circulating strain) levels for SWIM816 on D15 after study vaccination.

Cohorts 1: GMFR of SARS-CoV-2 Omicron (such as BA.5, BQ.1, XBB) and reference strain neutralizing.

antibody (other circulating strain) levels for SWIM816 on D15 after study vaccination.

Cohorts 1: % of participants with seroresponse to SWIM816 for GMTs of SARS-CoV-2 Omicron(such as BA.5, BQ.1, XBB) and reference strain neutralizing antibody (other circulating strain) levels on D15 after study vaccination.

Cohorts 2 (≥18 years ) Non-inferiority analysis: Geometric Mean Ratio (GMR) of SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB)-neutralizing antibody (other circulating strain) levels for SWIM816 to Pfizer Bivalent vaccine on D15 after study vaccination.

Endpoints:

Occurrence of local and systemic AEs reported within 7 days after study vaccination.

Occurrence of unsolicited AEs reported within 28 days after vaccination. Frequency, severity and relatedness of adverse events within 28 days after vaccination booster dose.

Endpoints:

Cohorts 1+2 : GMTs of Pseudovirus SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB) and reference strain neutralizing antibody levels for SWIM816 before and on D29, D91, D181 after study vaccination.

Cohorts 1+2 : GMFR of SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB) and reference strainneutralizingantibody levels for SWIM816 before and on D29, D91, D181 after study vaccination.

Cohorts 1: % of participants with seroresponse to SWIM816 for GMTs of SARS-CoV-2 Omicron(such as BA.5, BQ.1, XBB) and reference strain neutralizing antibody (other circulating strain) levels on D29, D91, D181 after study vaccination.

Cohorts 1 : GMTs and GMI of IgG profile at D01, D15, D29 , D91and D181 of each study group.

Cohorts 1: GMTs of Pseudovirus SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB) and reference strain neutralizing antibody levels for SWIM516 before and on D15, D29, D91, D181 after study vaccination.

Cohorts 1: GMFR of SARS-CoV-2 Omicron (such as BA.5, BQ.1,XBB) and reference strain neutralizing antibody levels for SW-BIC-213 before and on D15, D181 after study vaccination.

Endpoints:

Serious AEs (SAEs), AEs leading to withdrawal and AEs of special interest (AESIs) within 180 days.

Endpoints:

Occurrence of confirmed symptomatic cases during the study period. Number of confirmed SARS-CoV-2 symptomatic cases; Severity of confirmed cases of SARS-CoV-2 infection(WHO scale). Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subsets on D8 and Day 15 [ Time Frame: Day 8 and Day 15 after the study vaccination .]

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years old when signing ICF.
2. Participants who were previously vaccinated with 2/3 doses of COVID-19 vaccine, with or without previously diagnosed with COVID-19. The interval between the date of last dose and the date of this study vaccination should be 6 to 24 months.
3. Those who have not been infected with the novel coronavirus or have been infected for more than 3 months.
4. The participant and/or his legally acceptable representative can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial.
5. The participant and/or his legally acceptable representative have the ability to read, understand, and fill in record cards.
6. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment.
7. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

1. Presence of fever within 3 days before the study vaccination;
2. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or other disease corresponding use of immunosuppressants;
3. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
4. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
5. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.
6. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
7. Those who are tested positive for HIV in terms of serology.
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
12. Participants who received other investigational drugs or vaccines within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart f ailure, acute sore throat,hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
15. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
16. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
17. Those who plan to donate ovum or sperms during the study period;
18. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
19. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase II :Immunogenicity | 15 days after study vaccination
  GMTs of SARS-CoV-2 Omicron and related strain neutralizing antibody levels for SWIM816.
Phase II :Immunogenicity | 14 days post dose
  To demonstrate the non- inferiority of neutralizing antibody response in terms of geometric mean titers (GMT) of COVID-19 mRNA vaccine(SWIM816) compare with mRNA COVID-19 vaccine(Pfizer Bivalent vaccine) 14 days post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mayfong Mayxay, doctor, Principal Investigator — National Ethics Committee for Health Research(NECHR)

IPD SHARING:
Plan to Share IPD: No